CLINICAL TRIAL: NCT00608855
Title: Percutaneous US and CT-guided Cryoablation of Painful Metastases Involving Bone: A Feasibility Study
Brief Title: Percutaneous Cryoablation in Treating Patients With Painful Bone Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: MC03C3; MAYO-MC03C3
Record Dates: First submitted 2008-02-01; First posted 2008-02-06 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: bone metastases; pain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Cryosurgery; Analgesia

INTERVENTIONS:
Other: questionnaire administration
Procedure: cryosurgery
Procedure: pain therapy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Percutaneous cryoablation may help relieve pain caused by bone metastases.

PURPOSE: This clinical trial is studying the side effects and how well percutaneous cryoablation works in treating patients with painful bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* To confirm the safety of percutaneous cryoablation in the palliative treatment of patients with painful bone metastases.
* To determine the benefits of cryoablation of painful bone metastases by assessing pain intensity using a standardized Cleeland Brief Pain Inventory (BPI) and quality of life using a standardized SF-8 both before and after treatment.
* To determine the secondary benefits of cryoablation of painful bone metastases by assessing change in analgesic use following therapy.
* To determine the level of anesthesia required for cryoablation with a baseline level of conscious sedation planned for each treatment.

OUTLINE: This is a multicenter study.

Patients undergo percutaneous cryoablation to one or two sites of metastatic disease using the Endocare Cryocare system. Patients with a good initial response to treatment (≥ 2 decrease in pain intensity rating on the Brief Pain Inventory) who develop recurrent pain at the same site or a new painful site ≥ 1 month after initial treatment may undergo one additional cryoablation treatment.

Patients complete pain and quality of life questionnaires periodically.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic solid tumor involving or abutting bone (index lesion)

  * If the nature of the metastatic disease has been previously documented, index lesion to be treated does not require further documentation (i.e., biopsy)
* Pain either refractory to standard care (chemotherapy, radiotherapy, surgery, or analgesics) or patient is considered a poor candidate for conventional therapies

  * Radiation oncology consult is required if the patient is considered clinically to be a candidate for conventional palliative radiotherapy
  * Surgical oncology consult is required if the patient is considered clinically to be a candidate for conventional surgical treatment or is considered at risk for complications resulting from potential fracture
* Initial pain score ≥ 4 on a scale of 0-10 for the question "Please rate your pain by circling the one number that best describes your pain at its worst in the past 24 hours" on the Cleeland Brief Pain Inventory

  * Pain from ≤ 2 sites of metastatic disease
* No lesions with evidence for impending fracture involving a weight-bearing bone (> 50% loss of cortical bone at the site)

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 2 months
* Platelet count ≥ 75,000/mm³
* ANC > 1,500/mm³ (for patients who have recently been treated with chemotherapy)
* INR ≤ 1.2
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior radiotherapy
* More than 3 weeks since initiation of a new chemotherapy regimen, including bisphosphonates
* More than 7 days since prior antiplatelet medications or clopidogrel
* More than 3 days since prior acetylsalicylic acid (aspirin), ibuprofen, or other NSAIDs
* No prior treatment of the portion of a lesion within 0.5 cm of the spinal cord or brain, within 0.5 cm of a large abdominal vessel such as the aorta or inferior vena cava, or within 1 cm of bowel or bladder
* No prior radiofrequency ablation for pain palliation of the same lesion
* No concurrent regular or low molecular weight heparin or other anticoagulants

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Average difference in pre- and post-treatment worst pain score in a 24-hour period at week 8

SECONDARY OUTCOMES:
Average difference in pre- and post-treatment worst pain score in a 24-hour period, average pain score, and pain relief score at 6, 12, and 24 months
Average amount of pain per patient over the observation period as represented by the area under the curve (AUC) constructed from weekly pain scores on a visual-analogue scale using a score of 0-10
Percentage of patients who are able to reduce analgesic medications

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Callstrom, MD, PhD, Study Chair — Mayo Clinic
Locations (10):
- United States (10):
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University School of Medicine, Providence, Rhode Island
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin